CLINICAL TRIAL: NCT05157373
Title: The Effect of Androgen Receptor Polymorphism on Endometrial Cancer Development, Progression, and Outcome
Brief Title: The Effect of Androgen Receptor Polymorphism on Endometrial Cancer
Acronym: AREC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Nicosia (Other)
Responsible Party: Principal Investigator, Dionysis Vaidakis, Clinical Assistant Professor, University of Nicosia
Other Study IDs: DV001
Record Dates: First submitted 2021-05-08; First posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Androgen Receptor Abnormal; Endometrial Disorder
Keywords: Androgen Receptor; CAG; Receptor polymorphism
MeSH Terms: conditions — Bulbo-Spinal Atrophy, X-Linked

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — endometrial tissue and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Patients with any type of endometrial cancer
  Interventions: Diagnostic Test: Endometrial sampling and Peripheral blood collection; Behavioral: FSFI Scale
- Group 2: Patients with hyperplastic endometrial lesion (all type of endometrial hyperplasia and endometrial polyps). In this group will be included the breast cancer survivors under tamoxifen.
  Interventions: Diagnostic Test: Endometrial sampling and Peripheral blood collection; Behavioral: FSFI Scale
- Control group: A random sample of women without any endometrial pathology.
  Interventions: Diagnostic Test: Endometrial sampling and Peripheral blood collection; Behavioral: FSFI Scale

INTERVENTIONS:
Diagnostic Test: Endometrial sampling and Peripheral blood collection — The endometrial biopsy will be performed with a pipette. The pipelle will be inserted gently through the cervix and into the uterus. The pipelle procedure takes approximately one minute and involves gently moving the pipelle back and forth to obtain a sample. Then 10cc of peripheral blood will be collected.
Behavioral: FSFI Scale — The participants will fill up the Female Sexual Function Index (FSFI) questionnaire.
  The FSFI is a 19-item self-report questionnaire designed to measure sexual functioning in women. It assesses six domains of sexual function: sexual desire, sexual arousal, lubrication, orgasm, satisfaction, and pain (i.e., pain associated with vaginal penetration).

SUMMARY:
Endometrial tissue is a hormonal-dependent tissue in both pre- and postmenopausal period. The endometrial cells are expressing receptors for all sex hormones, mainly for estrogen, progesterone and androgens. The proper response of the endometrial cells on hormones is crucial for a well-balanced fluctuation of endometrial tissue. If, for any reason, these responses are altered, this may lead to benign or malignant lesions.

The androgens, through their receptors, decrease the proliferation of the endometrial cells. After menopause, the number of androgens receptors (ARs) increases in proportion to estrogen receptors and this may lead to endometrial atrophy. If the functionality of ARs is decreased, the effect of estrogen increases and this may possibly lead to endometrial hyperplasia or to endometrial cancer. The AR gene is located on the X chromosome and consists of 8 exons. Genetic research has shown that on exon 1, there is an area of trinucleotide Cytosine- Adenosine- Guanin (CAG) repeats which controls the functionality of the receptor. The more CAG repeats, the less responsive the receptor.

The goal of this research is to study the AR gene polymorphism and particularly the number of CAG repeats on exon 1, in patients with known endometrial pathology (benign and malignant). The results will be compared with a random sample of the general population without endometrial pathology.

DETAILED DESCRIPTION:
The role of CAG repeats on the AR is well established in degenerative neurological diseases in prostate and breast cancer, but the corresponding role in endometrial benign or malignant lesions is not well studied. It seems that there is a gap in the international literature since the results of the published studies are conflicting. A meta-analysis of 51 studies published by Qin et al. in 2017, suggested that the carriers of short polymorphic CAG repeats might increase the risk of prostate cancer, and could be used as a potential detecting marker. Another meta-analysis of 17 studies concluded that the longest CAG repeats increase the risk of breast cancer. Both those cancers are testosterone dependent and the higher the testosterone serum levels, the greater the cancer risk. Among women, the highest testosterone serum levels are observed in polycystic ovarian syndrome (PCOS) patients. A study published in 2020 concluded that the risk of PCOS is associated with the inheritance of ARs with shorter CAG repeats.Even though a meta-analysis of 11 studies demonstrate no evident association between the CAG length in AR gene and PCOS risk, the CAG length appears to be positively associated with higher testosterone levels. However, larger scale case-control studies are needed to validate the results. The rationale of the present study is to contribute to the literature by correlating the number of CAG repeats on AR with specific endometrial benign or malignant lesions. This may result in a better understanding of the nature of endometrial lesions and the development of specific clinical interventions.

The goal of this research is to study the AR gene polymorphism and particularly the number of CAG repeats on exon 1, in patients with known endometrial pathology (benign and malignant). The results will be compared with a random sample of the general population without endometrial pathology.

Impact on science, economy and society Adrenal receptor gene polymorphism seems to be related to many clinical conditions. Studying the AR gene polymorphism in relation to endometrial functionality will provide better understanding of the physiology of endometrial tissue function, the natural progression of endometrial lesions, as well as the potential of recurrence of those lesions after treatment. This may lead to the modification of therapeutic interventions and to the development of screening tests in high-risk populations.

Compliance Statement This study will be conducted in full accordance with all applicable research policies and procedures and all applicable laws and regulations. All episodes of noncompliance will be documented. The investigators will perform the study in accordance with this protocol, will obtain consent and assent, and will report unanticipated problems involving risks to subjects. Collection, recording, and reporting of data will be accurate and will ensure the privacy, health, and welfare of research subjects during and after the study.

ELIGIBILITY:
Inclusion Criteria

1. Women with histologically diagnosed primary endometrial cancer. All stages of endometrial cancer patients can be included in this group.
2. Women with the following endometrial lesion:

   1. Endometrial polyps
   2. Endometrial hyperplasia with and without atypia
   3. Endometrial hyperplasia after tamoxifen
3. Women with histologically proven normal endometrium

Exclusion Criteria:

1. Women with metastatic cancer in endometrium
2. Women with triple negative breast cancer
3. Women unable to consent

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study will be conducted at 2 investigative sites in Greece and Cyprus. Recruitment will stop when approximately 150 patients are enrolled.
  The study will be conducted at UNIC and will include patients from Anticancer Oncological Hospital of Athens ''Saint Savvas Hospital'' and from the researchers' private practices (control group and patients with benign endometrial lesions). All patients meeting the inclusion criteria below will be identified.
  Up to 150 selected cases from among eligible patients will be enrolled in the study protocol.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
The length of CAG repeats on exon 1 of AR gene and the relation to endometrial cancer vs control group | Day 1
  DNA analysis is required for the CAG repeat testing procedure. The DNA will be isolated from venous white blood cells and from endometrial cells. The high-molecular-weight DNA will then be analysed by polymerase chain reaction (PCR) amplification protocols, the exon 1 of the androgen receptor gene will be located and the number of CAG repeats will be recorded. If PCR is not sufficient to determine the exact number of replicates per case, the nucleotide sequence of the PCR products will be determined.
The length of CAG repeats on exon 1 of AR gene and the relation to benign lesions of the endometrium vs control group | Day 1
  DNA analysis is required for the CAG repeat testing procedure. The DNA will be isolated from venous white blood cells and from endometrial cells. The high-molecular-weight DNA will then be analyzed by PCR amplification protocols, the exon 1 of the androgen receptor gene will be located and the number of CAG repeats will be recorded. If PCR is not sufficient to determine the exact number of replicates per case, the nucleotide sequence of the PCR products will be determined.
The length of CAG repeats on exon 1 of AR gene as a predictive factor for endometrial lesions | Day 1
  DNA analysis is required for the CAG repeat testing procedure. The DNA will be isolated from venous white blood cells and from endometrial cells. The high-molecular-weight DNA will then be analyzed by PCR amplification protocols, the exon 1 of the androgen receptor gene will be located and the number of CAG repeats will be recorded. If PCR is not sufficient to determine the exact number of replicates per case, the nucleotide sequence of the PCR products will be determined.

SECONDARY OUTCOMES:
The length of CAG repeats on exon 1 of AR gene and the relation to endometrial cancer stage at diagnosis among group 1 patients | Day 1
  DNA analysis is required for the CAG repeat testing procedure. The DNA will be isolated from venous white blood cells and from endometrial cells. The high-molecular-weight DNA will then be analyzed by PCR amplification protocols, the exon 1 of the androgen receptor gene will be located and the number of CAG repeats will be recorded. If PCR is not sufficient to determine the exact number of replicates per case, the nucleotide sequence of the PCR products will be determined.
The length of CAG repeats on exon 1 of AR gene and the relation to endometrial cancer type among group 1 patients | Day 1
  DNA analysis is required for the CAG repeat testing procedure. The DNA will be isolated from venous white blood cells and from endometrial cells. The high-molecular-weight DNA will then be analyzed by PCR amplification protocols, the exon 1 of the androgen receptor gene will be located and the number of CAG repeats will be recorded. If PCR is not sufficient to determine the exact number of replicates per case, the nucleotide sequence of the PCR products will be determined.
The length of CAG repeats on exon 1 of AR gene and the relation to sexual function of the participants. | Day 1
  DNA analysis is required for the CAG repeat testing procedure. The DNA will be isolated from venous white blood cells and from endometrial cells. The high-molecular-weight DNA will then be analyzed by PCR amplification protocols, the exon 1 of the androgen receptor gene will be located and the number of CAG repeats will be recorded. If PCR is not sufficient to determine the exact number of replicates per case, the nucleotide sequence of the PCR products will be determined.
  The finding will be correlated with the answers of the participants in FSFI scale (Female Sexual Functioning Index )

CONTACTS AND LOCATIONS:
Overall Officials: Maria Chryssi, MSh, Principal Investigator — Anticancer oncological hospital of Athens "St Savvas'; Dionysios Vaidakis, MD,PhD., Study Director — Department of Life & Health Sciences, University of Nicosia; Adonis Ioannides, MD,PhD., Study Chair — Department of Life & Health Sciences, University of Nicosia

REFERENCES:
- [Result] Chuffa LG, Lupi-Junior LA, Costa AB, Amorim JP, Seiva FR. The role of sex hormones and steroid receptors on female reproductive cancers. Steroids. 2017 Feb;118:93-108. doi: 10.1016/j.steroids.2016.12.011. Epub 2016 Dec 29. PMID 28041951
- [Result] Sanderson PA, Critchley HO, Williams AR, Arends MJ, Saunders PT. New concepts for an old problem: the diagnosis of endometrial hyperplasia. Hum Reprod Update. 2017 Mar 1;23(2):232-254. doi: 10.1093/humupd/dmw042. PMID 27920066
- [Result] Maybin JA, Critchley HO. Menstrual physiology: implications for endometrial pathology and beyond. Hum Reprod Update. 2015 Nov-Dec;21(6):748-61. doi: 10.1093/humupd/dmv038. Epub 2015 Aug 7. PMID 26253932
- [Result] Zitzmann M, Nieschlag E. The CAG repeat polymorphism within the androgen receptor gene and maleness. Int J Androl. 2003 Apr;26(2):76-83. doi: 10.1046/j.1365-2605.2003.00393.x. PMID 12641825
- [Result] Qin Z, Li X, Han P, Zheng Y, Liu H, Tang J, Yang C, Zhang J, Wang K, Qi X, Tang M, Wang W, Zhang W. Association between polymorphic CAG repeat lengths in the androgen receptor gene and susceptibility to prostate cancer: A systematic review and meta-analysis. Medicine (Baltimore). 2017 Jun;96(25):e7258. doi: 10.1097/MD.0000000000007258. PMID 28640128
- [Result] Mao Q, Qiu M, Dong G, Xia W, Zhang S, Xu Y, Wang J, Rong Y, Xu L, Jiang F. CAG repeat polymorphisms in the androgen receptor and breast cancer risk in women: a meta-analysis of 17 studies. Onco Targets Ther. 2015 Aug 13;8:2111-20. doi: 10.2147/OTT.S85130. eCollection 2015. PMID 26316780
- [Result] Student S, Hejmo T, Poterala-Hejmo A, Lesniak A, Buldak R. Anti-androgen hormonal therapy for cancer and other diseases. Eur J Pharmacol. 2020 Jan 5;866:172783. doi: 10.1016/j.ejphar.2019.172783. Epub 2019 Nov 8. PMID 31712062
- [Result] Rosenfield RL, Ehrmann DA. The Pathogenesis of Polycystic Ovary Syndrome (PCOS): The Hypothesis of PCOS as Functional Ovarian Hyperandrogenism Revisited. Endocr Rev. 2016 Oct;37(5):467-520. doi: 10.1210/er.2015-1104. Epub 2016 Jul 26. PMID 27459230
- [Result] Polat S, Karaburgu S, Unluhizarci K, Dundar M, Ozkul Y, Arslan YK, Karaca Z, Kelestimur F. The role of androgen receptor CAG repeat polymorphism in androgen excess disorder and idiopathic hirsutism. J Endocrinol Invest. 2020 Sep;43(9):1271-1281. doi: 10.1007/s40618-020-01215-7. Epub 2020 Mar 12. PMID 32166698
- [Result] Baculescu N. The role of androgen receptor activity mediated by the CAG repeat polymorphism in the pathogenesis of PCOS. J Med Life. 2013 Mar 15;6(1):18-25. Epub 2013 Mar 25. PMID 23599814
- [Result] Zhang T, Liang W, Fang M, Yu J, Ni Y, Li Z. Association of the CAG repeat polymorphisms in androgen receptor gene with polycystic ovary syndrome: a systemic review and meta-analysis. Gene. 2013 Jul 25;524(2):161-7. doi: 10.1016/j.gene.2013.04.040. Epub 2013 Apr 26. PMID 23628801